CLINICAL TRIAL: NCT00972660
Title: A Phase II, Randomized Study to Evaluate the Safety and Efficacy of Ex-Vivo Cultured Allogenic Mesenchymal Stem Cells For the Treatment of Extensive Chronic Graft Versus Host Disease
Brief Title: Safety and Efficacy Study of Allogenic Mesenchymal Stem Cells to Treat Extensive Chronic Graft Versus Host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDREC.[2009]008
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2010-05

CONDITIONS: Graft Versus Host Disease
Keywords: Mesenchymal stem cell; Efficacy; Safety
MeSH Terms: conditions — Graft vs Host Disease | interventions — Methylprednisolone; Cyclosporine; Tacrolimus; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): Patients with newly diagnosed extensive cGVHD receive prednisone and cyclosporine or tacrolimus.
  Patients with refractory extensive cGVHD receive primary treatment (eg,prednisone and cyclosporine or tacrolimus, or plus mycophenolate mofetil, or methotrexate.)
  Interventions: Drug: Prednisone and cyclosporine or primary therapies
- Mesenchymal stem cell (MSC) (Experimental): Patients with newly diagnosed extensive cGVHD receive MSC plus prednisone and cyclosporine or tacrolimus.
  Patients with refractory extensive cGVHD receive MSC plus their primary immunosuppressive treatment (eg. prednisone + cyclosporine or tacrolimus, or plus mycophenolate mofetil, or plus methotrexate.)
  Interventions: Biological: Mesenchymal stem cell (MSC)

INTERVENTIONS:
Biological: Mesenchymal stem cell (MSC) — Experimental:Mesenchymal stem cell(MSC). Patients with newly diagnosed extensive cGVHD: prednisone 1mg/kg + cyclosporine or tacrolimus and MSC 2×1,000,000 MSC/kg, IV twice a week for the first two weeks and weekly for the following two weeks(6 doses totally).
  Refractory extensive cGVHD: receive primary treatment (prednisone + cyclosporine or tacrolimus, or plus mycophenolate mofetil, or plus methotrexate ) and MSC2×1,000,000 MSC/kg, IV twice a week for the first two weeks and weekly for the following two weeks(6 doses totally).
  Other Names: Medrol; Sandimmun Neoral; FK506,prograf; Cellcept; MTX
  Arms: Mesenchymal stem cell (MSC)
Drug: Prednisone and cyclosporine or primary therapies — Patients with newly diagnosed extensive cGVHD: prednisone 1mg/kg + cyclosporine or tacrolimus
  Patients with refractory extensive cGVHD: primary treatment (eg.prednisone 1mg/kg + cyclosporine or tacrolimus,or plus mycophenolate mofetil, or methotrexate.)
  Other Names: Medral; Sandimmun Neoral; FK506,Prograf; Cellcept,MMF; MTX
  Arms: Control group

SUMMARY:
Study Design: Treatment, Randomized, Open Label, Parallel Assignment,Safety/Efficacy Study.

The purpose of this study is to evaluate the safety and efficacy of mesenchymal stem cells (MSC) expanded ex-vivo infusion for the treatment of patients who have developed a newly diagnosed extensive or refractory chronic graft versus host disease (chronic GVHD) to the usual therapeutic measures.

DETAILED DESCRIPTION:
Chronic graft-versus-host disease (GVHD) is one of the main limitations to successful allogeneic hematopoietic stem cell transplantation (HSCT), and has a substantial impact not only on survival but also on the quality of life of otherwise cancer-free patients. Half of the patients undergoing a HLA-identical allografts who survive beyond 100 days may require long-term immunosuppressive treatment for extensive chronic GVHD, often for more than 2 years. More than one-third of patients with chronic GVHD do not respond to first-line therapy, which often involves combinations of corticosteroids and a calcineurin inhibitor. There is no standard second-line or salvage therapy for these patients and they have a poor outcome.

Mesenchymal stem cells (MSCs) are multipotent non-hematopoietic stem cells that can differentiate into various lineages and have been used to repair injured tissues. Recently, MSCs have also shown unique immunomodulatory properties ex-vivo, including inhibition of T-cell proliferation after stimulation by allo-antigens and mitogens, and prevention of the activity of cytotoxic T cells.MSCs have been used for the prophylaxis of acute GVHD and for the treatment of patients with steroid-refractory acute GVHD,but rarely have been used for extensive chronic GVHD.

Development of new therapeutic agents and strategies to rescue patients with extensive chronic GVHD would provide a significant benefit in an area of unmet medical need.

In this study, a single center randomized, non blinded Phase II clinical trial is proposed to study the safety and efficacy of mesenchymal stem cells (MSC) in the management of extensive chronic GVHD newly or refractory to the usual therapeutic measures.

Expanded MSC will be infused at a dose of 2 million cells/kg twice a week for 2 weeks and weekly for the following two weeks (six doses totally)in patients based first-line therapy (steroid plus cyclosporin A ) or their primary immunosuppressive therapies.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from patient and donor.
* Any patient who has undergone allogeneic stem cell transplantation with extensive chronic GVHD.
* Have not received additional agent for cGVHD within 3 months.
* Expected life is more than 90 days.
* Adequate pulmonary function with no evidence of chronic obstructive or severe restrictive pulmonary disease.
* Adequate cardiac function with no evidence of uncontrolled high blood pressure,congestive heart failure, angina pectoris, acute myocardial infarction within 6 months prior to the process.

Exclusion Criteria:

* Invasive fungal disease.
* Active cytomegalovirus (CMV)/Epstein-Barr virus(EBV)/varicella disease).
* Patient is with a history of hypersensitivity to bovine products.
* Relapsed malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2009-09; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The total Response rate defined as patients with complete and partial response. | Within the first 3 months (plus or minus 7 days) after randomization

SECONDARY OUTCOMES:
Overall Survival | Randomization until death or two years post last subject last treatment visit (or clinical cutoff)
Events Free Survival | Randomization until death or two years post last subject last treatment visit (or clinical cutoff)
The percentage of patients who can taper or discontinue the immunosuppressive agents | Randomization untill two years post the last subject last treatment visit (or clinical cutoff)
Serum cytokine levels and lymphocyte subsets in patients with chronic GVHD | Achieve best response within the first 3 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Xin Du, MD.PhD., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China